CLINICAL TRIAL: NCT03349398
Title: Uncut Roux-en-Y vs Roux-en-Y Reconstruction After Distal Gastrectomy for Gastric Cancer
Brief Title: Uncut Roux-en-Y vs Roux-en-Y
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jilin University (Other)
Responsible Party: Principal Investigator, Dong Yang, Assisted Investigator, Jilin University
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 130000
Record Dates: First submitted 2017-11-12; First posted 2017-11-21 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Uncut Roux-en-Y; Roux-en-Y; Gastric Cancer
Keywords: Uncut Roux-en-Y; Roux-en-Y
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the group of Roux-en-Y (Active Comparator)
  Interventions: Procedure: Roux-en-Y reconstruction
- the group of Uncut Roux-en-Y (Experimental)
  Interventions: Procedure: Uncut Roux-en-Y reconstruction

INTERVENTIONS:
Procedure: Uncut Roux-en-Y reconstruction — Uncut Roux-en-Y Reconstruction All surgical procedures will be performed by the single surgery team ,which is leaded by professor Wang Quan. Uncut Roux-en-Y construction will be used in this group.
  Arms: the group of Uncut Roux-en-Y
Procedure: Roux-en-Y reconstruction — Roux-en-Y Reconstruction All surgical procedures will be performed by the single surgery team ,which is leaded by professor Wang Quan. Roux-en-Y construction will be used in this group.
  Arms: the group of Roux-en-Y

SUMMARY:
Uncut Roux-en-Y vs Roux-en-Y reconstruction after distal gastrectomy for gastric cancer

DETAILED DESCRIPTION:
To search which is the better reconstructions by comparing and analyzing the advantages and disadvantages between Uncut Roux-en-Y and Roux-en-Y reconstructions after laparoscopy-assisted distal gastrectomy for gastric cancer.

Method: It's a prospective study including all patients underwent laparoscopy-assisted distal gastrectomy (LADG) in the First Hospital of Jilin University. All surgical procedures will be performed by the single surgery team, which is leaded by professor Wang Quan. The reconstruction method will be selected randomly from Uncut Roux-en-Y and Roux-en-Y anastomosis preoperatively without distinct indications. All clinical data, operation data, perioperative complications and related physiological indexes after surgery will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of distal gastric cancer
* underwent laparoscopy-assisted distal gastrectomy

Exclusion Criteria:

* have simultaneously other cancer
* have severe systemic inflammatory disease ,serious illness such as diabetes, chronic lung diseases
* have upper gastrointestinal surgery
* can't bear the gastric tube
* the period is too late or the tumor is too large to carry on a laparoscopy assisted radical distal gastrectomy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2017-11-10 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-06-02 (Estimated)

PRIMARY OUTCOMES:
the incidence of Roux stasis syndrome | 3 month after surgery
  the incidence of Roux stasis syndrome after Roux-en-Y reach an incidence of over 30% which involve nausea, vomiting, and abdominal distension. So the incidence of both reconstructions should be compared.

SECONDARY OUTCOMES:
the incidence of other complications after operation | one month after surgery
the quility of life according to the RGB standards | 12 month after surgery
  the RGB standards in Terms of Gastritis, Bile Reflux, and Gastric Residue

CONTACTS AND LOCATIONS:
Overall Officials: Quan Wang, Doctor, Study Director — The First Hospital of Jilin University
Locations (1):
- the First Hospital of Jilin University, Ch’ang-ch’un, Jilin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cai Z, Mu M, Ma Q, Liu C, Jiang Z, Liu B, Ji G, Zhang B. Uncut Roux-en-Y reconstruction after distal gastrectomy for gastric cancer. Cochrane Database Syst Rev. 2024 Feb 29;2(2):CD015014. doi: 10.1002/14651858.CD015014.pub2. PMID 38421211